CLINICAL TRIAL: NCT01620502
Title: N-3 Polyunsaturated Fatty Acids in the Prevention and Treatment for IFN-induced Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Kuan-Pin, China Medical University Hospital, National Science and Technology Council, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NSC98-2628-B-039-020-MY3
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Major Depressive Episode
MeSH Terms: interventions — Fatty Acids, Omega-3; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- EPA 3.5 g/day (Active Comparator)
  Interventions: Dietary Supplement: Omega-3 fatty acids
- Placebo capsules (Placebo Comparator): oleic oil
  Interventions: Dietary Supplement: Omega-3 fatty acids
- DHA 1.75 g/day (Experimental): DHA 1.75 g/day
  Interventions: Dietary Supplement: Omega-3 fatty acids

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acids — A daily treatment of 5 identical capsules of EPA (3.5 g/d), DHA (1.75 g/d) or placebo (high oleic oil), in single or divided administration for 2 (Study 1) or 8 weeks (Study 2)
  Other Names: Omega-3 PUFAs or fish oil

SUMMARY:
The first part is a double-blind placebo-controlled trial to identify the effects of omega-3 polyunsaturated fatty acids (PUFAs) in prevention of IFN-induced depression. The second part is a double-blind trial to identify the antidepressant effects of omega-3 PUFAs in patients with IFN-induced depression.

DETAILED DESCRIPTION:
We have done a preliminary analysis in 63 HCV patients receiving IFN-α therapy enrolled in our current NSC project (NSC95-2320-B-039-037-MY3) and found that patients who later developed IFN-α-induced depression (case group, 21/63) had lower PUFA levels before starting IFN-α therapy than control group (p=0.024). In addition, there was a trend for a negative correlation (r=-0.224; p=0.078) between baseline DHA levels and the highest scores of BDI during IFN therapy in the whole group. These findings indicate that n-3 PUFAs might play a protective factor.

This 3-year proposal is divided into 2 clinical studies. In study 1, we aim to test the prophylactic effect of n-3 PUFAs (EPA: 3.5 g/d and DHA: 1.75 g/d versus placebo: high oleic oil) for IFN-α-induced sickness behaviour and depressive symptoms, in a two-week, double-blind, placebo-controlled trial of 152 patients with HCV starting IFN-α therapy. In study 2, we will test the antidepressant effect of n-3 PUFAs (EPA: 3.5 g/d and DHA: 1.75 g/d versus placebo: high oleic oil) on IFN-α-induced depression during IFN-α therapy, in an eight-week, double-blind, placebo-controlled trial in 80 HCV patients who have already developed depression.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be adult patients with chronic HCV, assessed by hepatologists and then referred for IFN-α therapy and have capacity and willingness to give written informed consent

Exclusion Criteria:

* Patients will be excluded if they have major depressive episode at assessment
* Any history of pre-existing psychotic disorders (e.g. schizophrenia or bipolar disorder)
* Alcohol or drug dependence within one year before entry into the study
* Seizure disorders and evidence of any unstable substantial coexisting medical conditions (e.g. cardiovascular, endocrine, haematological, renal, or neurological diseases)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2009-07; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with major depressive episode (for Study 1); Changes in Hamilton Depression Rating Scale (HDRS) (for Study 2) | Weeks 0 to 24

SECONDARY OUTCOMES:
Changes in Hamilton Depression Rating Scale (HDRS) (for Study 1); Response and remission rates (for Study 2) | Weeks 0 to 24

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Pin Su, MD PhD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Su KP, Lai HC, Yang HT, Su WP, Peng CY, Chang JP, Chang HC, Pariante CM. Omega-3 fatty acids in the prevention of interferon-alpha-induced depression: results from a randomized, controlled trial. Biol Psychiatry. 2014 Oct 1;76(7):559-66. doi: 10.1016/j.biopsych.2014.01.008. Epub 2014 Jan 24. PMID 24602409